CLINICAL TRIAL: NCT03842254
Title: Use of Erythropoietin to Expand Regulatory T Cells in Autoimmune Liver Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Mount Sinai Hospital, New York (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Josh Levitsky, Professor of Medicine and Surgery, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU00206077
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Autoimmune Hepatitis
MeSH Terms: conditions — Hepatitis, Autoimmune | interventions — Erythropoietin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single arm (Experimental): Single dose of erythropoietin 10,000 units to be administered subcutaneously at time of enrollment.
  Interventions: Drug: Erythropoietin

INTERVENTIONS:
Drug: Erythropoietin — Subcutaneous injection of erythropoietin 10,000 units

SUMMARY:
This study evaluates the effect of erythropoietin on the number and function of regulatory T cells in adults with autoimmune hepatitis. Participants will receive a single dose of erythropoietin, and then the investigators will collect blood at different time points for analysis of regulatory T cell number and function.

DETAILED DESCRIPTION:
There is data from the laboratory that erythropoietin helps stimulate regulatory T cells, a type of immune cell which is thought to combat autoimmunity, but this study will look at whether it does the same thing in adults with autoimmune hepatitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autoimmune liver diseases (autoimmune hepatitis, autoimmune cholangiopathy, or primary biliary cirrhosis or primary sclerosing cholangitis with hepatic autoimmune liver disease or overlap syndrome) confirmed on liver biopsy
* Use of immunosuppressive therapy (prednisone, azathioprine, 6-mercaptopurine, mycophenolate mofetil) for the treatment of the autoimmune liver disease
* Stable immunosuppression regimen at least 6 months prior to enrollment
* Ability to provide verbal and written informed consent

Exclusion Criteria:

* Diagnosis of decompensated cirrhosis (defined by presence of ascites, varices, encephalopathy)
* Hemoglobin above average normal value (15.7 g/dL in men, 13.8 g/dL in women)
* Alanine aminotransferase greater than 2 times upper limit of normal (33 IU/L in men and 25 IU/L in women)
* Uncontrolled hypertension with systolic blood pressure greater than or equal to 160 or diastolic blood pressure greater than or equal to 100
* End-stage renal disease on hemodialysis
* History of venous thromboembolism including deep vein thromboses or pulmonary emboli
* History of stroke
* History of heart failure
* History of seizure disorder
* History of significant cardiovascular disease including a history of myocardial infarction
* Active malignancy (untreated or undergoing therapy)
* History of pure red cell aplasia
* History of intolerance or allergy to erythropoietin
* Known hypersensitivity to mammalian cell-derived products
* Known hypersensitivity to human albumin
* Presence of vascular access
* Prior recipient of erythropoietin within 12 weeks of the study
* Patient unable to provide consent including infants, children, teenagers, prisoners, cognitively impaired adults
* Non-English speaking
* Pregnancy

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Change in number of regulatory T cells | At time of enrollment, then at 2 weeks, 4 weeks, and 12 weeks.
  Calculated relative to baseline collected at time of enrollment

SECONDARY OUTCOMES:
Change in number of effector T cells after a single dose of erythropoietin | At time of enrollment, then at 2 weeks, 4 weeks, and 12 weeks.
  Calculated relative to baseline collected at time of enrollment
Change in cytokine production by the T cells in response to ex vivo stimulation | At time of enrollment, then at 2 weeks, 4 weeks, and 12 weeks.
  Calculated relative to baseline collected at time of enrollment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Northwestern Medicine, Chicago, Illinois
  - Mount Sinai, New York, New York

REFERENCES:
- [Derived] McEachern E, Carroll AM, Fribourg M, Schiano TD, Hartzell S, Bin S, Cravedi P, Levitsky J. Erythropoietin administration expands regulatory T cells in patients with autoimmune hepatitis. J Autoimmun. 2021 May;119:102629. doi: 10.1016/j.jaut.2021.102629. Epub 2021 Mar 13. PMID 33721837